CLINICAL TRIAL: NCT05136976
Title: Rituximab Therapy in Anti-Myelin Associated Glycoprotein Patients With Characteristics of Good Responders:
Brief Title: Rituximab Therapy in Anti-Myelin Associated Glycoprotein Patients With Characteristics of Good Responders
Acronym: THERAMAG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19PH226; 2021-000009-25 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anti-MAG Neuropathy
Keywords: Neuropathy; Anti-MAG; Rituximab; I-RODS; placebo
MeSH Terms: interventions — Rituximab; Sodium Chloride; Premedication

STUDY DESIGN:
Intervention Model Description: The THERAMAG study is a French academic multicentre, randomized, double-blind trial sponsored by the University Hospital of Saint-Etienne, comparing rituximab infusion to placebo infusion in anti-MAG patients presumed as good clinical responders.
Who Masked: Participant, Investigator
Masking Description: The randomization will be performed by the pharmacy. The treatment group will not be mentioned to the clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patient with anti-MAG neuropathy will be included. They will randomized in placebo or Rituximab group.
  They will have the same premedications prior to rituximab or placebo infusions:
  * IV Dexchlorpheniramine Maleate IV: 10 mg
  * IV Methylprednisolone: 40 mg
  * PO Paracetamol : 1 gram
  Interventions: Drug: Placebo infusion; Drug: Premedications
- Rituximab (Active Comparator): Patient with anti-MAG neuropathy will be included. They will randomized in placebo or Rituximab group.
  They will have the same premedications prior to rituximab or placebo infusions:
  * IV Dexchlorpheniramine Maleate IV: 10 mg
  * IV Methylprednisolone: 40 mg
  * PO Paracetamol : 1 gram
  Interventions: Drug: Rituximab infusion; Drug: Premedications

INTERVENTIONS:
Drug: Rituximab infusion — 2 infusions of 1 gram of rituximab at a 2 week interval (day 1 followed by day 15).
  Other Names: Mabthera
  Arms: Rituximab
Drug: Placebo infusion — 2 infusions of placebo at a 2 week interval.
  Other Names: Sodium chloride (NaCl)
  Arms: Placebo
Drug: Premedications — Premedications prior to rituximab or placebo infusions:
  * IV Dexchlorpheniramine Maleate IV: 10 mg
  * IV Methylprednisolone: 40 mg
  * PO Paracetamol : 1 gram

SUMMARY:
Anti-MAG neuropathy is a progressively disabling orphan rare disorder due to a monoclonal immunoglobulin M(IgM) gammopathy displaying reactivity toward MAG, a glycoprotein of the peripheral nervous system. Its prevalence is around 1/100000 and to date, no treatment has proven efficacy in this disease, including rituximab in 2 Randomized Controlled Trails(RCTs).

DETAILED DESCRIPTION:
However these trials have included unselected anti-MAG patients and methodological issues have been raised.

In COFRAMAG study, the largest cohort worldwide of anti-MAG patients, predictors of clinical response to rituximab were identified through analysis of 92 treated patients: shorter disease duration and anti-MAG titre above 10000 BTU. Thus this study will focus on rituximab efficacy in a subset of patients with disease duration of less than 2 years and anti-MAG titre above 10000 Buhlmann Titer Units (BTU). The investigators selected Inflammatory Rasch-built Overall Disability Scale (I-RODS) as primary outcome measure because its responsiveness was proven higher than INCAT/ Overall Neuropathy Limitation Score (ONLS) scales to detect clinical meaningful changes in newly treated patients with inflammatory neuropathies.

ELIGIBILITY:
Inclusion Criteria:

* Disease duration of 5 years or less and documented clinical worsening (clinical or ENMG or disability) over the past 24 months
* IgM gammopathy, either MGUS or Waldenstrom Macroglobulinemia (WM)
* Demyelinating polyneuropathy according to European Federation of Neurological Societies/Peripheral Nerve Society guidelines for chronic inflammatory demyelinating polyneuropathy on nerve conduction studies.
* Anti-MAG titre of 10 000 BTU or more
* Total INCAT score of 1 point or more at baseline
* Absence of immunoglobulin treatment within 3 months prior to inclusion.
* Absence of immunosuppressive therapy within 6 months prior to inclusion, including steroid therapy of 2 months or more as part of the management of neuropathy.
* Negative β-human chorionic gonadotropin (HCG) in women of childbearing potential
* Women of childbearing potential must agree to use contraception for 365 days following administration of rituximab.

Exclusion Criteria:

* - Unable to give informed consent
* History of severe allergic or anaphylactic reaction to chimeric monoclonal antibody
* Hypersensitivity known to one of the compounds of polaramine or methylprednisolone
* Previous treatment with rituximab
* Diseases known to cause polyneuropathy (e.g. diabetes, uncontrolled thyroid disease, vitamin B1 or B12 deficiency, renal (GFR < 60ml ml/min/1,73 m2- Modification of Diet in Renal Disease (MDRD) formula) or liver disorder, myeloma, amyloidosis, cryoglobulinemia)
* Indication of specific immunosuppressive therapy for WM
* Significant uncontrolled disease at baseline such as cardiovascular (including cardiac arrhythmia), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine or gastrointestinal or any other significant disease that may prevent patient from participating in the study
* Congestive heart failure (NYHA III or IV)
* Known active bacterial, viral, fungal mycobacterial infection
* History or known presence of recurrent or chronic infection (e.g. viral hepatitis, HIV syphilis, tuberculosis).
* History of cancer, including solid tumors and haematological malignancies (except basal cell and in situ squamous carcinoma of the skin, in situ carcinoma of the cervix of the uterus that have been excised and resolved, with documented clear margins on pathology)
* History of alcohol (more than two drinks a day for a woman, more than 4 glasses a day for a man [World Health Organization (WHO) definition]) or other drug abuse within 6 months prior to randomization
* History or currently active primary or secondary immunodeficiency
* White blood cell count < 1500/mm3 or platelet count < 75 000/mm3
* Angle closure glaucoma,
* Urinary retention related to urethroprostatic disorders,
* Uncontrolled psychotic disorders,
* Severe liver failure,
* Recent vaccination with live vaccines (<3months) and vaccination with live virus vaccines is not recommended during the overall study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
I-RODS score | Baseline and 12 months
  Clinical response defined as a 4 points (or more) change of I-RODS between baseline and 12 months.
  I-RODS is a 24-item patient-reported outcome measure which maximum score is 48. It is a linearly weighted scale that specifically captures activity and social participation limitations in patients with inflammatory neuropathies, including Monoclonal Gammopathy of Unknown Significance (MGUS) related polyneuropathies.

SECONDARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) disability score | Months: 0, 6, 12
  The INCAT (Inflammatory Neuropathy Cause and Treatment) disability score is a measure of activity limitation with minimum score at 0 and maximum at 10.
Six minute walk test | Months : 0, 6, 12
  Six minute walk test will be realized.
Timed 25- foot walk (FW) test | Months : 0, 6, 12
  The T25-FW is a quantitative test of mobility and performance of leg function based on a timed outward journey of 25 steps, and a timed return journey of 25 steps. The score for the T25-FW is the average of the two completed trials
9 hole peg test | Months : 0, 6, 12
  The nine hole peg test is a standardized, quantitative assessment used to measure finger dexterity. Scores are based on the time taken to complete the test activity, recorded in seconds
ElectroNeuroMyography (ENMG) | Months : 0, 6, 12
  An ENMG will be realized.
ENMG sensory sum score | Months : 0, 6, 12
  ENMG sensory sum score will be realized.
Score Motor unit number index (MUNIX) | Months : 0, 6, 12
  Score MUNIX will be realised.
Incidence of Treatment-Emergent Adverse Events of Rituximab | Months : 0, 6, 12
  Consideration of adverse effects of Rituximab
the anti-MAG antibody titre. | Months : 0, 6, 12
  To study the correlation between the clinical response and the evolution of the anti-MAG antibody titre.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure KAMINSKY, MD, Principal Investigator — CHU de Saint-Etienne
Locations (15):
- France (15):
  - CHU Brest - La cavale blanche, Brest
  - CHU Grenoble - La tronche, Grenoble
  - CHU Lille - Roger Salengro, Lille
  - CHU Limoges - Dupuytren, Limoges
  - HCL lyon, Lyon
  - CHU La Timone - APHM, Marseille
  - CHU Nancy- Hôpital central, Nancy
  - Hôtel-Dieu et Hôpital GR Laënnec - CHU Nantes, Nantes
  - CHU Nice - Pasteur, Nice
  - APHP Pitié Salpêtrière, Paris
  - APHP - Kremlin-Bicêtre, Paris
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU Strasbourg - Hautepierre, Strasbourg
  - CHU Toulouse - Pierre-Paul Riquet, Toulouse
  - CHU Tours - Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No